CLINICAL TRIAL: NCT06363981
Title: Multisite Repetitive Transcranial Magnetic Stimulation for Mood, Cognitive Impairment, Anhedonia and Disordered Sleep in Depressive Disorder
Brief Title: Multisite rTMS for Mood, Cognitive Impairment and Other Symptoms of Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jakub Antczak (Other)
Collaborators: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Sponsor-Investigator, Jakub Antczak, Clinical Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JagiellonianU72
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Unipolar Depression; Bipolar Disorder
Keywords: depression; repetitive transcranial magnetic stimulation; dorsolateral prefrontal cortex; dorsomedial prefrontal cortex; cognitive impairment; anhedonia; sleep disorders
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Depression; Cognitive Dysfunction; Anhedonia; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective, randomized, sham-controlled clinical trial in parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo intervention will be delivered with a programmable coil for magnetic stimulation, which can be switched by a third person between modes of active (therapeutic) and sham stimulation. In the sham-mode coil elicits similar sounds as in the active stimulation, but induces only negligible magnetic field.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMS over the left DLPFC and over the left DMPFC (Experimental): Active 10 Herz rTMS with intensity of 120% of the resting motor threshold recorded from the right first dorsal interosseus and the right abductor hallucis will be administered over the left DLPFC and over the left DMPFC respectively. Therapy will include 20 sessions (one session in each of 20 consecutive working days - four weeks in total). In every session ca 1500 magnetic pulses over the left DLPFC and ca 1500 over the left DMPFC will be elicited.
  Interventions: Device: Active rTMS over the left DLPFC and over the left DMPFC
- rTMS over the left DLPFC (Active Comparator): Active 10 Herz rTMS with intensity of 120% of the resting motor threshold recorded from the right first dorsal interosseus will be administered over the left DLPFC. Therapy will include 20 sessions (one session in each of 20 consecutive working days - four weeks in total). In every session 3000 magnetic pulses over the left DLPFC will be elicited.
  Interventions: Device: Active rTMS over the left DLPFC
- Sham rTMS (Sham Comparator): Sham 10 Herz rTMS will be administered over the left DLPFC. Therapy will include 20 sessions (one session in each of 20 consecutive working days - four weeks in total). In every session 3000 magnetic pulses over the left DLPFC or ca 1500 magnetic pulses over the left DLPFC and ca 1500 over the left DMPFC will be elicited. (rTMS protocol will be chosen randomly before the first session).
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS over the left DLPFC and over the left DMPFC — Active rTMS over the left DLPFC and over the left DMPFC to induce the long term potentiation of stimulated areas.
  Arms: rTMS over the left DLPFC and over the left DMPFC
Device: Active rTMS over the left DLPFC — Active rTMS over the left DLPFC to induce the long term potentiation of stimulated area.
  Arms: rTMS over the left DLPFC
Device: Sham rTMS — Sham rTMS over the left DLPFC or over the left DLPFC and over the left DMPFC for placebo.
  Arms: Sham rTMS

SUMMARY:
Depressed mood is the main symptom of depression, but other symptoms like cognitive impairment, anhedonia or sleep disorders may also contribute to patients suffering and are difficult to treat. rTMS is a relatively novel treatment option, whose therapeutic potential is still investigated and optimized. The aim of this study is to assess the effect of rTMS applied over two stimulation sites on cognitive impairment, anhedonia and sleep disorders in depression.

DETAILED DESCRIPTION:
Depression is one of the most common and disabling disorders, affecting approximately three hundred million people worldwide. Depressive mood is the main symptom, but other symptoms like cognitive impairment, anhedonia or sleep disorders contribute significantly to patients suffering, decrease quality of life and may even lead to suicide attempt. While modern pharmacotherapy can significantly improve symptoms in many patients, still one third of patients remains drug-resistant. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive method of inducing brain plasticity. Stimulation over the left and right dorsolateral prefrontal cortex (DLPFC) and possibly over several other areas can improve mood. Only few studies investigated the effect of rTMS on negative psychiatric symptoms, such as anhedonia, sleeplessness or cognitive impairment. In these trials, either the DLPFC or the dorsomedial prefrontal cortex (dmPFC) were stimulated and sometimes other areas such as the insular cortex. The aim of this study is to investigate if a stimulation over both sites (multi-site stimulation) has better therapeutic potential for depressed mood, cognitive impairment, anhedonia and sleep disorders than stimulation over DLPFC alone and placebo.

ELIGIBILITY:
Inclusion Criteria:

* severe or moderate depressive episode (according to international classification of diseases (ICD)-10) without psychotic symptoms at the time of inclusion
* Hamilton Depression Rating Scale between between 20 and 35 points at inclusion
* The score in the Athens Insomnia Scale eight or more
* The score of three or more points in items 4 and 21 of the Beck Depressions Inventory 2
* Complaining about problems with memory and concentration timely related with the onset of depression

Exclusion Criteria:

* Contraindications to transcranial magnetic stimulation, including ferromagnetic elements in head, pregnancy and epilepsy
* Psychotic symptoms at the time of inclusion
* Suicidal ideations and/or attempts within three months prior to inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory 2 | Before intervention - four weeks after finishing intervention.
  Inventory consisting of 21 items measuring cognitive, affective, somatic, and vegetative symptoms of depression. Each item is scored from 0 to 3, with a higher score denoting more severe depression. Items are related to the criteria from the Diagnostic and Statistical Manual of Mental Disorders-IV. The minimum value of the total score is 0 and the maximum is 63 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Froward digit span | Before intervention - four weeks after finishing intervention.
  A measure of verbal short term and working memory. Participant is asked to repeat the random series of numbers, which become longer along with every correctly repeated one. Test is finished after participant failed to respond correctly on three occasions. The number of correctly repeated series determines the final score, which is an integer representing the length of the largest passed sequence. The scores range from 3 to 9 with higher scores denoting better outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Language part of Addenbrooke's Cognitive Examination | Before intervention - four weeks after finishing intervention.
  A test to identify cognitive impairment in dementia. In the language part, participant is asked to complete a set commands such as "place the paper on top of the pencil"; to write grammatically-complete sentences; to repeat several words and proverbs; to name the objects shown in drawings, and answer questions and to read several mispronounced words. The number of correctly completed tasks is scored. The minimum value of the total score is 0 and the maximum (of the language part) is 26 with higher scores meaning better outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.

SECONDARY OUTCOMES:
Dimensional Anhedonia Rating Scale | Before intervention - four weeks after finishing intervention.
  A 17-item scale that measures desire, motivation, effort and consummatory pleasure across hedonic domains. In each item, participant chooses one of four statements describing his attitude towards a given activity. The minimum value of the total score is 0 and the maximum is 68 with higher scores meaning better outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Athens Insomnia Scale | Before intervention - four weeks after finishing intervention.
  An eight item scale. Each item is rated from 0 to 3 with higher scores representing more severe insomnia. Change from baseline score in the Athens Insomnia Scale to the measurement taken after finishing rTMS. The minimum value of the total score is 0 and the maximum is 24 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Pittsburgh Sleep Quality Index | Before intervention - four weeks after finishing intervention.
  Pittsburgh Sleep Quality Index (PSQI) is a questionnaire to identify sleep disturbances. It consists of a combination of Likert-type and open-ended questions, which are later converted to scaled scores. Scores for each question range from 0 to 3. The minimum value of the total score is 0 and the maximum is 21 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Epworth Sleepiness Scale | Before intervention - four weeks after finishing intervention.
  An eight-item scale. Each item refers to a situation such as driving a car or sitting quietly. The subject is asked to assess the chance of dosing in each situation, ranging from 0 (no chance) to 3 (dosing very likely). The minimum value of the total score is 0 and the maximum is 24 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Korzeniowski, MD, Principal Investigator — The Education of Research and Development Center, Babinski Clinical Hospital
Locations (1):
- The Education of Research and Development Center, Babinski Clinical Hospital, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Yes
Scans of scales, inventories and questionnaires will be available upon request sent per e-mail to: wojciech.korzen@gmail.com
Supporting Information: Study Protocol, SAP
Time Frame: December 2026 - December 2030
Access Criteria: For researchers in medical sciences and medical professional upon justification of their request.